CLINICAL TRIAL: NCT04588753
Title: Comparison of Active Isolated Stretch and Post Facilitation Stretch on Hamstring Flexibility in Trans-tibial Amputees
Brief Title: Active Isolated Stretch and Post Facilitation Stretch on Hamstring Flexibility in Trans-tibial Amputees.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00680 Tehmina Khan
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Amputation
Keywords: Trans-tibial Amputees; Isolated Stretch; Post Facilitation Stretch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Isolated Stretch (Active Comparator): active isolated stretching, strengthening exercises
  Interventions: Other: active isolated stretch
- Post Facilitation Stretch (Active Comparator): Post Facilitation Stretching, strengthening exercises
  Interventions: Other: Post Facilitation Stretch

INTERVENTIONS:
Other: active isolated stretch — Active Isolated Stretch (AIS);
  * The shortened hamstring muscle will be isolated.
  * The hamstring will be stretched.
  * This Stretches will be Repeated eight to 10 times.
  * Stretch will be hold for no more than two seconds.
  * Exhale on the stretch; inhale on the release. Other amputees training exercises;
  * weight-shifting
  * Dynamic balancing activities
  * Stool stepping
  * Braiding
  * Gait exercises
  * Climbing/descending the stairs
  Arms: Active Isolated Stretch
Other: Post Facilitation Stretch — Participants of this group will receive Post Facilitation Stretch (PFS);
  * The shortened hamstring muscle will be placed between a fully stretched and a fully relaxed state.
  * The patient will be asked to contract the hamstring using a maximum degree of effort for 5-10 seconds while the therapist will resists thepatients force.
  * The patient will be then asked to relax and release the effort, whereas the therapist will apply a rapid stretch to a new barrier and is held for 10 seconds.
  * The patient relaxes for approximately 20 seconds and the procedure will be repeated to five times (8) (18).
    2. Other amputees training exercises;
  * weight-shifting
  * Dynamic balancing activities
  * Stool stepping
  * Braiding
  * Gait exercises
  * Climbing/descending the stairs
  Arms: Post Facilitation Stretch

SUMMARY:
The aim of this study is to examine the effect of two techniques on hamstrings flexibility in trans-tibial amputees. Reduced flexibility can cause insufficiency at the workplace. Increasing flexibility is to decrease risk of injury, enhances performance and incorporate rehabilitation programs . Further studies are still needed in order to enhance patient rehabilitation protocol and anticipate the prosthetic process. Evidence based Physical therapy could be considered a valid support improving knee contractures in patients with trans-tibial amputation.This research provide an important addition to the evidence-based treatment intervention of physical therapy in amputees rehabilitation as no comparative study between Active Isolated Stretch and Post Facilitation Stretch on hamstring flexibility is done in trans-tibial Amputees.

DETAILED DESCRIPTION:
Trans-tibial amputation (Below-knee amputation) that involves removing the foot, ankle joint and distal tibia and fibula with related soft tissue structures . Amputations occurs due to variety of reasons including trauma, diseases, tumors, infections and congenital malformations .Traumatic amputations tend to occur in younger and active age and in Pakistani amputee population the majority 65-70% the cause of amputation is traumatic and 50-60% are Trans-tibial amputations. Several complications related to the amputation-prosthesis interface needs attention while managing amputees including joint full range of motion especially in the joint immediately proximal to the amputation site. The trans-tibial amputees are prone to develop flexion deformity of the knee . Normal active range of motion of the knee is 0° extension and 140° flexion. In many people after Tran's tibial amputation with a flexion deformity, active range of motion of the ipsilateral knee is reduced . The main cause of occurrence of flexion deformity of the knee is the muscle shortening and tightness especially the hamstrings muscles due to the long periods in a bending position or inactivity due to the illness or lack of exercise .

Muscle Energy Techniques are used for lengthening of the muscles and improve range of motion (ROM) in joints . Active Isolated Stretching (AIS) is a uniquely effective exercise system with the advantages of specificity, active initiation, Incremental assists, Gentle motion, Brief duration, Multiple repetitions and Deep breathing. To stretch the hamstring muscles by lifting the leg straight up, stay on the mid-sagittal plane (keep the legs parallel). If the leg rotates out to the side, you lose much of the hamstring stretch and start affecting other muscles instead . While In Post Facilitation Stretch technique the hypertonic and shortened muscle is placed between a fully stretched and a fully relaxed state. Contracture of hamstrings using a maximum degree of effort for 5-10 seconds while the therapist resists the force. After this relaxation is done and effort is released and the therapist applies a rapid stretch to a new barrier and is held for 15 seconds. The relaxation is for 20 seconds and the procedure is repeated between three to five times and five times more .

Study concluded that the AIS helps to restore the deteriorated flexibility of the muscles . In 2013 study concluded compare the Muscle Energy Techniques with static stretches' for increasing hamstring flexibility in post burn patients. Their results shows that Both treatment groups had highly significant gains in knee extension ROM after 5 and 8 days post stretching exercises. But MET had highly significant gains in knee extension ROM than static stretching after 8 days of treatments .

In 2014 studied the three groups of 60 male students of Semnan University of Medical Sciences having shortened hamstring muscles. The 1st group underwent the hold relax technique, 2nd group underwent static stretches' and the 3rd group with no interventions for 4 weeks and three times a week. Results were recorded with goniometer before and after the sessions. Their results showed that both methods have a significant effect on increasing the motion range of knee. But no significant difference was observed between the static stretch and hold-relax techniques .

In 2019 study reviewed 4 studies related to active isolated stretches' for knee extension who evaluated 53 subjects who performed knee extension stretches 4 times a week for 4 weeks. The increase in ROM was statistically significant after the 1st week of AIS and in static stretches after 2 to 4 weeks. The AIS increase in ROM was significantly greater than for the static stretch exercise. Another study studied 30 subjects and their results showed that both modes of stretching significantly increased ROM, but AIS increased ROM significantly more than the static stretch exercise. Another study evaluated 30 subjects and reported that only the AIS significantly increased ROM. study reported on 30 subjects concluded that AIS increased ROM more than 11% versus the 8% by static stretch but the difference was not statistically significant .

ELIGIBILITY:
Inclusion Criteria:

* Unilateral Trans-tibial amputees.
* Amputees having short hamstring (>15- 30 degrees loss of knee extension)
* Patients with traumatic cause of amputation.
* Patients that are mentaly stable.
* Patients having no other physical problems than amputation.
* Patient aged between 15 and 30 years.
* 1 year post amputation and ambulatory with a prosthesis.
* Both male and female patients

Exclusion Criteria:

* Amputees other than trans-tibial amputees.
* Patients having other cause of amputation than traumatic.
* Requiring intervention before the amputation

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension Test (AKE) | 2 weeks
  used to measure hamstring flexibility. The subject be asked to lie in supine position with the non-tested limb and the pelvis will be strapped to the plinth for stabilization. The tested leg will be positioned in 90 degrees of hip flexion and the knee flexed. Hip flexion will be maintained through the use of a crossbar to maintain the proper position of hip and thigh. A full circle universal goniometer will be used to measure the angle of knee ROM. The fulcrum of the goniometer will be centered over the lateral condyle of the femur with the fixed arm secured along the femur using the greater trochanter as a reference. The movable arm will be aligned with the lower leg using the lateral malleolus as a reference. Subject will be asked to actively extend the tested knee as far as possible until a mild stretch sensation is felt. The procedure will be repeated 3 times and the average will be taken for analysis. Amputees having short hamstring (>15- 30 degrees loss of knee extension)

CONTACTS AND LOCATIONS:
Overall Officials: Shafaq Shahid, MSPT(OMPT), Principal Investigator — Riphah International University
Locations (1):
- PIPOS Rehabilitation Services Program, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jabeen N, Malik S. Prevalence and pattern of traumatic limb amputations in female population of Bhimber District, Azad Jammu and Kashmir, Pakistan. Pak J Med Sci. 2015 Jan-Feb;31(1):54-9. doi: 10.12669/pjms.311.6423. PMID 25878614
- [Background] Kwan MK, Penafort R, Saw A. Treatment for flexion contracture of the knee during Ilizarov reconstruction of tibia with passive knee extension splint. Med J Malaysia. 2004 Dec;59 Suppl F:39-41. PMID 15941159
- [Background] Ghazali MF, Abd Razak NA, Abu Osman NA, Gholizadeh H. Awareness, potential factors, and post-amputation care of stump flexion contractures among transtibial amputees. Turk J Phys Med Rehabil. 2018 Jul 12;64(3):268-276. doi: 10.5606/tftrd.2018.1668. eCollection 2018 Sep. PMID 31453521
- [Background] Yigiter K, Sener G, Erbahceci F, Bayar K, Ulger OG, Akdogan S. A comparison of traditional prosthetic training versus proprioceptive neuromuscular facilitation resistive gait training with trans-femoral amputees. Prosthet Orthot Int. 2002 Dec;26(3):213-7. doi: 10.1080/03093640208726650. PMID 12562068
- [Background] Wrisley DM, Marchetti GF, Kuharsky DK, Whitney SL. Reliability, internal consistency, and validity of data obtained with the functional gait assessment. Phys Ther. 2004 Oct;84(10):906-18. PMID 15449976
- [Background] Page P. Current concepts in muscle stretching for exercise and rehabilitation. Int J Sports Phys Ther. 2012 Feb;7(1):109-19. PMID 22319684